CLINICAL TRIAL: NCT06007326
Title: A Multicentre, Retrospective Study of Clinical Characteristics and Long-term Outcomes of Patients With Brucellosis
Status: Completed | Type: Observational
Sponsor: Qin Ning (Other)
Responsible Party: Sponsor-Investigator, Qin Ning, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: REBEL
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Brucellosis
MeSH Terms: conditions — Brucellosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a multicenter, retrospective clinical study, in patients with brucellosis, to analyze the clinical characteristics, complications, and the impact of different treatment options on long-term prognosis of patients with brucellosis. All hospitalized patients diagnosed with brucellosis between 2016 and 2021 were included from the electronic medical record systems of eight centers, collecting demographics, hospitalization information, clinical information, laboratories, imaging studies, treatment regimens, and disease outcome and other information.

ELIGIBILITY:
Inclusion Criteria:

* Age and gender are not limited;
* Discharged patients diagnosed with brucellosis
* Specific reference to the People's Republic of China's health industry standard "Diagnosis for brucellosis" (WS269-2019) diagnosed as a patient with brucellosis, that is, the patient meets a suspected or clinically diagnosed case and passes the confirmatory test mentioned below at the same time Either to prove:

  1. Brucella is isolated from any pathological material culture such as blood, bone marrow, other body fluids and excreta of patients.
  2. The test tube agglutination test (SAT) titer is 1:100++ and above, or the patient's course of disease lasts for more than one year and still has clinical symptoms, and the titer is 1:50++ and above.
  3. Complement fixation test (CFT) titer is 1:10++ and above.
  4. Anti-human immunoglobulin test (Coomb's) titer is 1:400++ and above.
* Volunteer to join this study.

Exclusion Criteria:

* History of severe lumbar spine trauma before the diagnosis of brucellosis;
* Have undergone lumbosacral surgery before the diagnosis of brucellosis;
* Scoliosis;
* Currently participating in clinical trials of other drugs or medical devices;
* The researchers think it is not suitable for inclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients diagnosed with Brucellosis from 8 centers in Hubei Province, China.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics | 2 year
  The electronic medical record system was used to collect patients' symptoms from baseline (admission) to 24 months, including initial symptoms, constitutional symptoms and signs [fever (maximum temperature, duration), hyperhidrosis, muscle/joint soreness, fatigue, hepatomegaly, splenomegaly, testicular enlargement, oophoritis, lymphadenopathy (location and size), others].
Complication rate | 2 year
  Electronic medical record system was used to collect the complications of patients from baseline (admission) to 24 months, and the incidence of complications within 2 years was calculated.
  Complications include osteoarticular system (sacroiliitis, spondylitis, peripheral arthritis, osteomyelitis, bone destruction, etc.) that may be related to brucellosis, Genitourinary system (orchitis, epididymitis, oophoritis, glomerulonephritis, renal abscess, etc.), central nervous system (peripheral neuropathy, meningoencephalitis, mental symptoms, cranial nerves, chorea, etc.), skin (maculopapular rash, Cyst, Stevens-Johnson syndrome, etc.), respiratory system (pleural effusion, pneumonia, etc.), blood system (leukocyte increase or decrease, platelet deficiency, etc.), cardiovascular system (endocarditis, vasculitis, myocarditis wait). Diagnostic tests for complications include laboratory tests (blood routine, etc.), echocardiography, imaging tests (X-ray, ultrasound, high-resolution CT)

SECONDARY OUTCOMES:
Survival rate | 1 year,2 years
  The 1-year survival rate and 2-year survival rate were calculated.
Disease outcome (cured, improved, not cured, progress, relapse, death) | 2 year
  The electronic medical record system was used to collect the disease outcomes of patients from baseline (admission) to 24 months.
Etiological characteristics (B.melitensis [1, 2, 3 subtypes], B.abortus[1-9 subtypes], B.suis [1-5 subtypes], B.canis) | 2 year
  Etiologic characteristics were collected from baseline (admission) through 24 months with the use of an electronic medical record system. The distribution of pathogens was analyzed, and the relationship between different pathogenic characteristics and long-term prognosis (disease outcome) was evaluated.
Number of patients with severe brucellosis (ICU number) | 2 year
  The electronic medical record system was used to collect the proportion of patients admitted to ICU from baseline (admission) to 24 months, and the proportion of patients admitted to ICU was calculated.
antimicrobial therapy | 2 year
  The electronic medical record system was used to collect the treatment options of patients from baseline (admission) to 24 months, and the impact of different treatment options on prognosis (disease outcome) was evaluated.
Hospital costs | 2 year
  The electronic medical record system was used to collect the hospitalization expenses of patients, and the average hospitalization cost was calculated.

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Guangshui First Peoples Hospital, Guangshui, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - People's Hospital of Luotian County, Huanggang, Hubei
  - People's Hospital of Macheng city Affiliated Hospital of Hubei Univerciy of science and technology, Macheng, Hubei
  - Qianjiang Central Hospital, Qianjiang, Hubei
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - Yichang Third Peoples Hospital, Yichang, Hubei